CLINICAL TRIAL: NCT06587503
Title: EbolaCov: A Phase IV, Single-centre, Single-blinded, Randomized Controlled Trial to Assess Safety and Immunogenicity of rVSVΔG-ZEBOV-GP Vaccination When Dosed Concurrent With mRNA COVID-19 Vaccine Booster Doses in Healthy African Adults
Brief Title: Safety and Immunogenicity of rVSVΔG-ZEBOV-GP Vaccination When Dosed Concurrently With mRNA COVID-19 Vaccine Booster Doses
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Project San Francisco (Unknown); Rwanda Biomedical Centre (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EbolaCov; PACTR202407764378004 (Registry Identifier: Pan African Clinical Trials Registry)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Ebola Virus Disease; COVID-19
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; COVID-19 | interventions — BNT162 Vaccine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Receive an intramuscular injection of a placebo concurrently with a dose of rVSV∆G-ZEBOV-GP vaccine
  Interventions: Biological: 1mL saline solution; Biological: rVSV∆G-ZEBOV-GP
- Concurrent vaccination (Experimental): Receive an intramuscular dose of BioNTech - Pfizer COVID-19 concurrently with a dose of rVSV∆G-ZEBOV-GP vaccine
  Interventions: Biological: BioNTech - Pfizer COVID-19 vaccine; Biological: rVSV∆G-ZEBOV-GP

INTERVENTIONS:
Biological: BioNTech - Pfizer COVID-19 vaccine — Vaccine for protection from COVID-19
  Other Names: Cominarty
  Arms: Concurrent vaccination
Biological: 1mL saline solution — Placebo
  Other Names: rVSV∆G-ZEBOV-GP
  Arms: Placebo
Biological: rVSV∆G-ZEBOV-GP — Vaccine for protection from Zaire Ebola virus
  Other Names: Ervebo

SUMMARY:
Concurrent vaccination scheduling for key target populations in Rwanda, such as healthcare workers, may confer significant advantages in the provision of vaccine coverage to several infectious diseases. This is a phase IV vaccine trial that looks to establish if two licenced vaccines, the rVSVΔG-ZEBOV-GP vaccine for protection against Ebola virus and messenger ribonucleic acid (mRNA) COVID vaccine for protection against SARS-CoV-2 virus, given concurrently to self selected healthy adult volunteers confers an acceptable safety profile and immunogenicity response.

DETAILED DESCRIPTION:
Vaccines for the prevention of severe disease caused by Ebola virus and SARS-CoV-2 virus are routinely offered to adults at higher risk of exposure in African settings. For protection from Ebola virus, the main target populations are epidemiologically-identified and include healthcare workers, refugees, and people living in outbreak zones. These target populations are also routinely offered vaccines for other vaccine-preventable diseases. However, there are currently no data on whether the co-administration of rVSVΔG-ZEBOV-GP with other vaccines has an acceptable profile of reactogenicity and antigen-specific immunogenicity, and concomitant use of rVSVΔG-ZEBOV-GP with other vaccines is not recommended. Clinical trial data on the co-administration of rVSVΔG-ZEBOV-GP with other vaccines prioritised for the same population, and especially in the context of a new era in mRNA vaccine technology, would have significant relevance to how protection to more than one disease can be provided at a single visit to a vaccination clinic. This, in turn, has the potential to improve vaccine coverage and improve the efficiency of vaccine policy and logistics, as well as being the first step evaluation in the evaluation of Vesicular stomatitis virus-vectored vaccine technology with lipid-enveloped mRNA platforms that are going to be increasingly used in other formulations against other/future infectious diseases targets.

There are no preliminary data in this first-of-kind study.

The advent of the SARS-CoV-2 virus and COVID-19 pandemic signalled the accelerated development of lipid-nanoparticle mRNA vaccine technology with great success. The mRNA platform is highly adaptable to new disease targets, including cancer and infectious diseases pathogens, and a multitude of vaccine candidates are currently in development for outstanding global health priorities that have eluded pre-pandemic technologies. However, there remains very little known about using mRNA technologies in combination with, or concurrent to, other vaccine technologies and whether there are any adverse signals associated with safety or antigen-specific immune response/protection. Earlier trials have focussed on using SARS-CoV-2 mRNA vaccines in combination with adjuvant-protein vaccines for seasonal influenza (and herpes-zoster virus, in setup) and have reported favourable safety and humoral immune responses that has resulted in recommended concurrent vaccine dose administration into the annual seasonal vaccination schedule of UK nationals. These study data have significantly supported public confidence in accepting two licenced vaccines at the same time and significant efficiency gains in vaccine coverage and public protection. The concurrent administration of mRNA vaccines with attenuated or replication-incompetent viral-vectored vaccines has not, to our knowledge, been assessed although many trials reported favourable safety and immunogenicity with heterologous combinations of these vaccine platforms for protection against COVID-19. Since existing mRNA COVID-19 vaccines and new mRNA constructs against other infectious diseases are expected to become routine immunisations for key members of the population, such as healthcare workers and older adults, research is needed to inform whether concurrent or co-administration with other vaccines are possible. For African populations, the risk of disease outbreaks from Ebola remains high and the future use of rVSVΔG-ZEBOV-GP is expected, along with other measures, to mitigate the risks to healthcare workers and the wider public. Assessing the safety and immunogenicity of rVSVΔG-ZEBOV-GP vaccine in the context of expected gains in public confidence and policy implementation with co-administration with mRNA vaccine technologies is a major subject of interest for African populations and preparedness for future disease outbreaks.

This is a single-centre, randomized, single-blinded, vaccine safety and immunogenicity study in healthy adults living in Rwanda. The EbolaCov trial aims to inform whether the Ebola vaccine rVSVΔG-ZEBOV-GP can be administered concurrent to a BioNTech - Pfizer COVID-19 booster dose without an unacceptable increase in reactogenicity and/or loss of humoral immunogenicity to Ebola vaccine antigen.

The investigators aim to primarily recruit participants who are current healthcare workers, although the study will be open all eligible members of the public. Participants of both genders aged 18-50 years who are in good health and who are able to provide written informed consent, will be eligible for inclusion in this study. The recruitment target is recruit 72 participants who will be randomised in a 1:1 ratio to one of two groups.

There will be four study visits over 6 months. Participants will be monitored for any reactions and other adverse events for 7 days after each immunisation via self reported e-diary, and for significant adverse events throughout the study.

The geometric mean titre (GMT) and antigen-specific antibody titre will be measured by glycoprotein-enzyme-linked immunosorbent assay at baseline, 28-days and 180-days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between ages 18-50 years, who are able and willing to provide written informed consent and will comply with the study requirements.
* Already completed a primary course of COVID-19 immunisation (any World Health Organisation approved primary immunisation course is acceptable).

Exclusion Criteria:

* Unwilling or unable to provide written informed consent to take part
* Unwilling or unable to comply with study procedures
* Previously received an Ebola vaccine or previous exposure to Ebola virus (including serological and clinical diagnoses, irrespective of viral strain)
* Not received a primary course of COVID-19 immunisation
* History of any suspected or confirmed disorder of the immune system that, in the opinion of the Investigators, might impair the results of the study
* Use of immunosuppressant medication within the past 6 months (excluding topical steroids or oral steroid courses lasting <7 days)
* Current diagnosis or treatment of cancer (unless non-melanomatous skin cancer)
* Have a bleeding disorder deemed significant by study doctor
* Pregnant or breast-feeding females
* Able to avoid close contact with vulnerable individuals, including via high-risk blood and bodily fluids for 6 weeks following vaccination to reduce the risk of transmission to vulnerable individuals (e.g. immuno-compromised individuals, individuals receiving immunosuppressive therapy, pregnant or breast-feeding women, children <1 year of age).
* Unable to prevent contact of their blood or bodily fluids with farm animals in the 6 weeks following vaccination
* Plan to donate blood in the 6 weeks following vaccination
* Hypersensitivity to any active substances, excipients, or rice protein.
* History of anaphylaxis to any component of vaccine formulation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events in the seven days following vaccination | Day 7 post vaccination
  Rates of severe treatment related adverse events within one week of concurrent vaccine dose administration, compared to when rVSVΔG-ZEBOV-GP vaccine is given alone.
Day 28 serum anti-glycoprotein (GP) antibody responses | Day 28 post vaccination
  Serum anti-glycoprotein (GP) antibody responses 28-days after concurrent vaccine dose administration, compared to when rVSVΔG-ZEBOV-GP vaccine is given alone

SECONDARY OUTCOMES:
Day 28 and day 180 serum anti-GP and serum SARS-CoV-2 anti-Spike protein specific geometric mean titres | Day 180 post vaccination
  Longitudinal assessment of serum anti-GP and serum SARS-CoV-2 anti-Spike protein specific geometric mean titres after concurrent vaccine dose administration, compared to when rVSVΔG-ZEBOV-GP vaccine is given alone.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Green, PhD, Principal Investigator — University of Birmingham

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are not openly available to protect the confidentiality of study participants. Fully anonymised data are, however, available from the authors upon reasonable request and with permission from Merck Sharp & Dohme, if required.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting immediately after article publication and the data will be made accessible for up to 5 years. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a methodologically sound research proposal. Data must be required to achieve the aims in the approved proposal. Data requests should be directed to c.a.green.2@bham.ac.uk.

REFERENCES:
- [Derived] Gokani K, Taylor A, Packham A, Musabyimana JP, Shema H, Mutabaruka A, Roche S, Takwoingi Y, Umuhoza C, Nyombayire J, Muvunyi C, Green C. Safety and immunogenicity of rVSVDeltaG-ZEBOV-GP vaccination when dosed concurrent with mRNA COVID-19 vaccine booster doses in healthy African adults (EbolaCov): protocol for a phase IV, single-centre, single-blinded, randomised controlled trial. BMJ Open. 2025 Sep 21;15(9):e102898. doi: 10.1136/bmjopen-2025-102898. PMID 40976661